CLINICAL TRIAL: NCT03076515
Title: A Prospective, Randomized, Double-blind, Sham Controlled Multi-center Clinical Trial, Migraine Headache Treatment With Nerivio Migra Neurostimulation Device
Brief Title: Migraine Treatment With Nerivio Migra Neurostimulation Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was prematurely stop based on DMC recommendation
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCH_002
Record Dates: First submitted 2017-03-07; First posted 2017-03-10 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2020-10

CONDITIONS: Acute Migraine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Nerivio Migra active (Active Comparator): This arm will use the active device for acute treatment of migraine at the migraine symptoms onset. the device will be applied on the upper arm and controlled by a dedicated smartphone application.
  Interventions: Device: Nerivio Migra neurostimulation
- Nerivio Migra placebo (Sham Comparator): This arm will use the sham device for acute treatment of migraine at the migraine symptoms onset. the device will be applied on the upper arm and controlled by a dedicated smartphone application.
  Interventions: Device: Sham Nerivio Migra

INTERVENTIONS:
Device: Nerivio Migra neurostimulation — transcutaneous electrical stimulation
  Arms: Nerivio Migra active
Device: Sham Nerivio Migra — electrical stimulation- shame mode
  Arms: Nerivio Migra placebo

SUMMARY:
This is a prospective, randomized, double-blind, sham controlled multi-center trial. Ratio between treatment and control groups will be 1:1, stratified by center and use of preventive medications.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, sham controlled multi-center clinical trial "Migraine Treatment with Nerivio Migra electro stimulation device". The study will enroll up to 248 patients diagnosed with migraine with and without aura, per the inclusion and exclusion criteria. These patients will be individually and randomly assigned to either treatment group or control group. For sham control, short electrical pulses of amplitude range similar to that of the treatment programs will be administered at very low frequency (0.1-0.5 Hz). The rationale underlying selection of sham control settings is that, on the one hand, pulses are perceivable and the user is able to manipulate their intensity similarly to the case of treatment programs, while, on the other hand, no clinically relevant treatment is delivered, based on existing knowledge of parameters range of electro stimulation treatmentsץ

Following successful screening, enrollment interview and signing of informed consent, participants will be provided with an active Nerivio Migra or identically looking sham device and trained to perform treatment and provide feedback via the smartphone application. Ratio between treatment and control groups will be 1:1.

Baseline information including mean frequency and severity of migraine attacks, occurrence of other headaches, presence of ICHD-3 diagnostic criteria for migraine with and without aura and use of preventive and rescue medications will be recorded.

Investigational devices will be programmed in active or sham mode with a 1:1 ratio, in order to achieve the desired ratio between active and control groups sizes.

Stage One. In stage one (roll-in phase) recruited participants will be reporting their migraine attacks per ICHD-3 diagnostic criteria, including presence of aura, using an electronic migraine diary installed on their smartphones. Duration of this phase is one month.

Participants that will report less than 2 or more than 8 migraine attacks during the roll-in period will be excluded from the treatment phase.

Stage Two. This will be the parallel arm treatment stage. Participants will be instructed to activate the device at onset of a qualifying migraine attack and manually adjust stimulation intensity to a level within the pre-defined range where it is well perceived but not painful. A qualifying migraine attack shall be preceded by at least 48 hours of freedom from headache. Patients will be requested to refrain from use of rescue medications prior to and during the first two hours after treatment with the device, and if they can not comply with this, record their use of rescue medications (migraine specific drugs or other medications or therapies that may be used to treat pain, from a pre-specified list) in the mobile application.

Via the smartphone application, each participant will be asked to rate his/her migraine pain level three times using Pain Grades Scale (0 - no pain, 1- mild pain, 2- moderate pain, 3 - severe pain): (1) upon starting the treatment, (2) two hours after start of treatment, (3) 48 hours after start of attack. At the start of each treatment, participants will be also asked to provide time elapsed from start of migraine attack to start of the treatment. Participants will be also asked to provide feedback regarding their use of medication (migraine specific drugs or other medications or therapies that may be used to treat pain, from a pre-specified list), presence of nausea, photophobia and phonophobia, and treatment perception. After providing feedback at two hours after start of treatment and in case of pain recurrence, participants will be allowed to re-treat the attack using Migra device.

Adverse events will be reported. Duration of study participation for each patient will be up to three months, determined by one month of the roll-in stage followed treatment of four qualifying attacks over the course of two months (whichever is achieved first).

Post study questionnaire will include patient global impression of change, blinding and usability assessments.

Stage Three. This part will include open label extended treatment. Following the completion of the study by all subjects and the return of all study devices, subjects will be offered a 2-month period of using active device, at no cost.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18-75 years old.
2. Patient meeting the ICHD-3 diagnostic criteria for migraine with and without aura.
3. Patients reporting 2-8 migraine attacks per month.
4. Patient must be able and willing to comply with the protocol.
5. Patient must be able and willing to provide written informed consent.
6. Male or non-pregnant / non-lactating female (NOTE: Females of child bearing potential must have a negative pregnancy test) and must be willing to use adequate contraceptive means during the study

Exclusion Criteria:

1. Has other significant pain problem that in the opinion of the investigator may confound the study assessments
2. Is currently implanted with an electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagus nerve neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator cochlear implant, Sphenopalatine ganglion stimulator or Occipital nerve stimulator).
3. Known uncontrolled epilepsy.
4. Use of Cannabis including medical use.
5. Has chronic migraine (more than 15 headache days per month).
6. Changed usage or dosage of migraine preventive medications in the last two months
7. Has undergone nerve block (occipital or other) in the head or neck within the last 2 weeks.
8. Is participating in any other clinical study. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Grosberg, MD, Principal Investigator — Hartford Healthcare Headache Center
Locations (8):
- United States (4):
  - MedStar - Georgetown University Hospital, Washington D.C., District of Columbia
  - Albany Medical College, Albany, New York
  - Hartford Healthcare Headache Center, Hartford, New York
  - Northwell Health, Inc, New York, New York
- Israel (4):
  - Hillel Yaffe Medical Center, Hadera
  - Herzeliya medical Center, Herzliya
  - Maccabi Healthcare neurology clinics, Kfar Saba
  - Western Galilee Medical Center, Nahariya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nerivio Migra Active | Nerivio Migra Placebo
Started | 58 | 62
Completed | 33 | 33
Not Completed | 25 | 29
Not completed — DMC decision based on interim analysis | 25 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nerivio Migra Active | Nerivio Migra Placebo | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (12.9) | 42.3 (12.7) | 44.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 33 | 33 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Migraine attacks per month [Mean (Standard Deviation); unit: number of migraine attacks per month] | 4.0 (1.2) | 3.9 (1.3) | 4.0 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pain Relief 2 Hours Post Treatment
Description: Percentage of participants reporting pain relief from pain (pain reduction from 3 or 2 to 1 or 0 or pain reduction from 1 to 0) 2 hours post treatment without rescue medications in at least 50% of treated attacks
Time Frame: 2 hours post treatment
Measure: Number; unit: percentage of responded participants
Groups:
- Nerivio Migra Active: Subjects received an active form of Nerivio Migra neurostimulation device
- Nerivio Migra Placebo: Subjects received a Sham form of Nerivio Migra: neurostimulation device
Arm/Group | Nerivio Migra Active | Nerivio Migra Placebo
Number analyzed (Participants) | 33 | 33
percentage of responded participants | 36.3 | 27.2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Nerivio Migra Active | Nerivio Migra Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

LIMITATIONS AND CAVEATS:
Study was terminated following an interim analysis based on 25% of the target study sample size (performed on September 3rd, 2017). Interim analysis showed major protocol deviation in both study arms, both in treatment start time (from onset of migraine attack) and use of concomitant medications, technically considered as failure. Hence, The DMC decision was to terminate the study due to futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT03076515/Prot_SAP_000.pdf